CLINICAL TRIAL: NCT04850820
Title: Impact of Amino Acids to Enhance Anabolism After Home-based Exercise
Acronym: B2B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Iovate Health Sciences International Inc (Industry)
Responsible Party: Principal Investigator, Daniel Moore, Associate Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: B2B
Record Dates: First submitted 2021-04-17; First posted 2021-04-20 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Amino Acids, Essential; Metabolism; Exercise
Keywords: Home-based resistance exercise; Protein synthesis; Net protein balance; Protein breakdown; Essential amino acids; Branched-chain amino acids; Protein metabolism
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: In a randomized, counterbalanced order, participants will receive all treatments arms (essential amino acids, branched-chain amino acids, and placebo).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All investigators involved with the study, as well as participants, will be blinded to treatment conditions (double-blind design) until data analysis is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Novel essential amino acid supplementation (EAA+) (Experimental): Arm will investigate the effect of a novel essential amino acid-based formula (essential amino acids enriched with active botanical compounds; EAA+) developed by Iovate Health Sciences International Inc. on post-exercise anabolism. The formulation was recently granted a Natural Product Number (NPN: 80087022) and approved by the Natural and Non-prescription Health Products Directorate of Health Canada.
  Interventions: Dietary Supplement: Novel essential amino acid supplementation
- Branched-chain amino acid supplementation (BCAA) (Active Comparator): Arm will used a branched-chain amino acid supplement developed by Iovate Health Sciences International Inc. to compare with the experimental arm after exercise.
  Interventions: Dietary Supplement: Branched-chain amino acid supplementation (BCAA)
- Isocaloric carbohydrate supplementation (Placebo Comparator): Carbohydrate supplement that is isocaloric to the EAA+ supplement and designed to function as a placebo to the experimental arm after exercise.
  Interventions: Dietary Supplement: Isocaloric carbohydrate supplementation
- Rested control (Other): Carbohydrate supplement that is isocaloric to the EAA+ supplement but consumed at rest to serve as the baseline control
  Interventions: Dietary Supplement: Isocaloric carbohydrate supplementation

INTERVENTIONS:
Dietary Supplement: Novel essential amino acid supplementation — This intervention will determine the impact of EAA+ on markers of whole-body net protein balance, protein synthesis, and protein breakdown following home-based resistance exercise in a free-living setting.
  Arms: Novel essential amino acid supplementation (EAA+)
Dietary Supplement: Branched-chain amino acid supplementation (BCAA) — This intervention will determine the impact of the BCAA supplement (to be compared to EAA+) on markers of whole-body net protein balance, protein synthesis, and protein breakdown following home-based resistance exercise in a free-living setting.
  Arms: Branched-chain amino acid supplementation (BCAA)
Dietary Supplement: Isocaloric carbohydrate supplementation — This intervention will determine the impact of an isocaloric carbohydrate placebo supplement (to be compared to EAA+) on markers of whole-body net protein balance, protein synthesis, and protein breakdown following home-based resistance exercise in a free-living setting.
  Arms: Isocaloric carbohydrate supplementation; Rested control

SUMMARY:
An adequate quantity of lean body mass is vital for optimal health and performance, and is accrued when net protein balance (NPB) is positive. Amino acids are the building blocks of protein, and when consumed following resistance exercise, significantly improve NPB.

However, no study has investigated how a supplement of all of the essential amino acids (EAA) affects NPB following resistance exercise in a free-living, home-based setting, particularly when compared to a supplement of branched-chain amino acids (BCAA).

Therefore, the purpose of this study is to determine the impact of a novel EAA supplement on anabolism (e.g., NPB) as compared to BCAA and placebo supplements following home-based resistance exercise.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-35 years
* Recreationally active; currently performing structured exercise (e.g., running, weight lifting, team-sport activity) at least 2 days per week

Exclusion Criteria:

* Body Mass Index: >29.9kg/m^2
* Inability to perform physical activity as determined by the Physical Activity Readiness Questionnaire
* Inability to adhere to protocol guidelines (e.g., alcohol, habitual diet)
* Regular tobacco use
* Illicit drug use (e.g., growth hormone, testosterone)
* Diagnosed medical condition under the care of a physician
* Inability to abstain from supplements (e.g., protein, creatine, HMB, BCAA, phosphatidic acid) at least three weeks before and during trials
* Individuals on any medications known to affect protein metabolism (e.g., corticosteroids, non-steroidal anti-inflammatories, or prescription-strength acne medications)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Whole-body net leucine balance (umol/kg) | 5 hours/trial (four trials total)
  Used as a proxy of whole-body protein balance, and estimated by using [13C]leucine ingestion and breath/urine sample collection

SECONDARY OUTCOMES:
Urinary 3-methylhistidine (3-methylhistidine:creatinine ratio) | 5 hours/trial (four trials total)
  Used as a marker of muscle protein breakdown by measuring the 3-methylhistidine:creatinine ratio in the urine

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Moore, Principal Investigator — University of Toronto
Locations (1):
- Goldring Centre for High Performance Sport, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No